CLINICAL TRIAL: NCT01313468
Title: Effect of Aerobic Interval Training on NEAT in Sedentary Men
Brief Title: Interval Training and Resting Metabolism
Acronym: NEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010/1541
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Healthy Subjects
Keywords: NEAT; maximal oxygen uptake; stroke volume

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4 x 4 Interval (Experimental): 4 x 4 minutes of high intensity intervals at 90-95% of maximal heart rate separated by 3 minutes of active brakes in between at 70% of maximal heart rate.
  Interventions: Behavioral: 4 x 4 minutes Intervals
- 1 4 minutes interval (Experimental): 1 x 4 minutes intervals at 90-95% of HR max
  Interventions: Behavioral: 1 x 4 minute interval
- Moderate continuous Training (Experimental): 47 minutes of Moderate continuous Training
  Interventions: Behavioral: Moderate continuous Training

INTERVENTIONS:
Behavioral: 1 x 4 minute interval — 1 x 4 minutes of high intensity intervals at 90-95% of maximal heart rate
  Arms: 1 4 minutes interval
Behavioral: 4 x 4 minutes Intervals — 4 x 4 minutes of high intensity intervals at 90-95% of maximal heart rate separated by 3 minutes of active brakes in between at 70% of maximal heart rate.
  Arms: 4 x 4 Interval
Behavioral: Moderate continuous Training — 47 minutes of Moderate continuous Training
  Arms: Moderate continuous Training

SUMMARY:
It has been reported that obese individuals are seated 2 ½ hour more than lean individuals and that non exercise thermo genesis (NEAT) may vary with as much as 2000 Kcal/day between equal size people due to different occupational and leisure time activities. The primary aim of the study is to investigate if 10 weeks of exercise training increase NEAT in sedentary men.

Subject will be randomized to three different training intervention, with 3 exercise session each week for 10 weeks. NEAT will be measured using an activity sensor and recorded over a 7 day period both before and after training.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Age 18-50
* BMI 25-30 kg x m2
* No significant comorbidities
* Abel to exercise
* Not partaking in organized physical activity

Exclusion Criteria:

* Inability to exercise due to musculoskeletal conditions
* Known ischemic cardiovascular disease
* High daily physical and occupational activity levels

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
nonexercise activity thermogenesis | Baseline and 10 weeks
  NEAT Will be measured using an activity sensor. Physical activity is recorded over a 7 day period. The energy equivalent of each of these activities is determined. The time spent in each activity is then multiplied by equivalent for the activity. The values are then summed to derive an estimate of NEAT.

SECONDARY OUTCOMES:
Cardiopulmonary maximal oxygen uptake | Baseline and 10 weeks
  The secondary aims are to investigate the changes in maximal oxygen uptake, heart function, and body composition in response to interval training

CONTACTS AND LOCATIONS:
Overall Officials: Trine Karlsen, Principal Investigator — National Taiwan Normal University
Locations (1):
- NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zisko N, Stensvold D, Hordnes-Slagsvold K, Rognmo O, Nauman J, Wisloff U, Karlsen T. Effect of Change in VO2max on Daily Total Energy Expenditure in a Cohort of Norwegian Men: A Randomized Pilot Study. Open Cardiovasc Med J. 2015 Apr 30;9:50-7. doi: 10.2174/1874192401509010050. eCollection 2015. PMID 25969700